CLINICAL TRIAL: NCT03261050
Title: Target Engagement of a Novel Dissonance-Based Treatment for DSM-5 Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Stice, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH111782; 1R61MH111782 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorder
Keywords: Eating disorder; Counter attitudinal therapy; fMRI
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Project Treatment (Experimental): An 8-session group-delivered eating disorder treatment that seeks to reduce valuation of the thin ideal and eating disordered behaviors used to pursue this ideal.
  Interventions: Behavioral: Counter Attitudinal Therapy
- Interpersonal Psychotherapy (Active Comparator): An 8-session group-delivered eating disorder treatment that seeks to improve interpersonal functioning because this is theorized to maintain eating pathology.
  Interventions: Behavioral: Counter Attitudinal Therapy; Behavioral: Interpersonal Therapy

INTERVENTIONS:
Behavioral: Counter Attitudinal Therapy — 8 weekly 60 minute sessions of dissonance-based treatment wherein women with any eating disorder complete verbal, written, and behavioral activities.
Behavioral: Interpersonal Therapy — 8 weekly 60 minute sessions of interpersonal-based treatment wherein women with an eating disorder complete verbal, written, and behavioral activities.
  Arms: Interpersonal Psychotherapy

SUMMARY:
Most people with an eating disorder (ED) do not receive good treatment. The investigators have developed a new brief group treatment that is supposed to work by reducing how much women with an ED value the impossible thinness standard promoted by the media and how much they value/crave binge foods. The investigators want to test whether the treatment actually changes those two mechanisms using brain scan data, which is more objective than completing questionnaires and even interviews.

In the first phase of the study (R61), the investigators will compare women in the treatment versus those on a wait-list. If the investigators can show that the treatment "works" (does what the investigators think it does) compared to no active treatment (women will be allowed to seek and receive outside help but investigators will not provide it until after the wait-list), investigators will conduct the second phase of study (R33),where they will randomly assign women with an ED to either the new treatment or to a group treatment that represents what many college mental health clinics provide to their clients with ED.

DETAILED DESCRIPTION:
Only 3-20% of individuals with eating disorders (EDs) receive treatment, and those who do rarely receive evidence-based treatments because they are very intensive and costly, few clinicians deliver them, and they differ for the various EDs. These factors have hindered broad implementation of evidence-based treatments, implying that a brief frontline outpatient treatment for a range of EDs that could be easily, cheaply, and widely implemented would address a major public health problem. There is also limited experimental evidence regarding factors that maintain EDs and mechanisms of action for ED treatments. The investigators propose to conduct a project that translates basic persuasion research into clinical hypotheses and a novel treatment.

The investigators hypothesize that EDs are maintained by (1) excessive valuation of the thin beauty ideal, which prompts caloric restriction and other unhealthy weight control behaviors (vomiting, laxative use, excessive exercise) that increase binge eating risk, and (2) excessive valuation of high-calorie foods, which maintains binge eating. The investigators propose to evaluate a treatment that addresses these hypothesized maintenance processes. Two pilot trials evaluated a novel 8-session group dissonance-based treatment (Counter Attitudinal Therapy; CAT) wherein women with any ED appropriate for outpatient care completed activities in which they collectively discuss costs of pursuing the thin ideal and the ED behaviors in which they personally engage (unhealthy weight control behaviors and binge eating), which putatively creates dissonance about engaging in those particular behaviors that reduce valuation of the thin ideal and high-calorie binge foods.

During the COVID-19 shelter-at-home orders taking place at both research sites, the investigators will not measure in-person only outcomes including fMRI, ECG, computerized implicit associated tests, and height and weight measurements for all participants that have assessments during this order. The investigators will continue to conduct treatment groups that will be administered on a virtual platform.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 eating disorder
* Must have a primary care doctor

Exclusion Criteria:

* Non-English speakers
* BMI <75% ideal body weight
* Current acute suicidal ideation (defined as thoughts of a specific method or plan)
* Comorbid psychiatric disorder that would disrupt groups (e.g., bipolar disorder, substance misuse)
* Serious medical problems (e.g., diabetes)

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in occurrences of binge eating episodes using Eating Disorder Diagnostic Interview | Week 8; R33 also reviews at 6-month follow-up
  Interviewer assesses frequency in binge eating episodes
Change in occurrences of compensatory weight control behavior using Eating Disorder Diagnostic Interview | Week 8; R33 also reviews at 6-month follow-up
  Interviewer assesses frequency of compensatory weight control behaviors
Change in psychosocial impairment due to eating disorder symptoms using the Clinical Impairment Assessment Questionnaire | Week 8; R33 also reviews at 6-month follow-up
  Interviewer assesses change in psychosocial impairment

SECONDARY OUTCOMES:
Change in reward region of the brain using fMRI | Week 1 and Week 8
  Assess if CAT produces larger pre-post reductions in reward region in response to thin models and binge food (Not collected during COVID-19 shelter-at-home order)
Change in suicidal ideation/attempts using the Patient Health Questionnaire version 9 (PHQ-9) | Weeks 2, 4 and 6
  Assess if there are any changes in suicide ideation/attempts
Change in negative affect using the Positive Affect and Negative Affect Scale-Revised | Weeks 2, 4, and 6
  Assess if there are any changes in negative affect
Change in body dissatisfaction using the Body Dissatisfaction Scale | Weeks 2, 4 and 6
  Assess if there are any changes in body dissatisfaction
Change in food addiction using the Yale Food Addiction Scale version 2.0 | Weeks 2, 4, and 6
  Assess if there are any changes in food addiction (Only collected during R61 phase)
Change in valuation of thin ideal using the Thin Ideal Valuation Scale | Weeks 2, 4, 6, and 8; R33 also reviews at 6-month follow-up
  Assess if there are any changes in valuation of the thin beauty ideal
Change in dietary restraint using the 10-item Dutch Restrained Eating Scale | Week 8; R33 also reviews at 6-month follow-up
  Assess if there are any changes in dietary restraint
Change in implicit associations of binge foods, thin models, and eating disorder behavior words | Week 8; R33 also reviews at 6-month follow-up
  Three implicit association tasks will assess response to binge foods, thin models, and eating disorder behavior words at pre- and post-test (Not collected during COVID-19 shelter-at-home order)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Oregon Research Institute, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared via the National Database for Clinical Trials Related to Mental Illness (NDCT), which is part of the NIMH Data Archive (NDA). All data, with the exception of video recordings of the participants in treatment, will be provided.
Supporting Information: Study Protocol, CSR
Time Frame: Descriptive/raw data will be submitted while the study is ongoing (every 6 months). Analyzed data will be submitted either when results are published or after the completion of the award period, whichever comes first.

REFERENCES:
- [Result] Stice E, Yokum S, Rohde P, Shaw H, Gau JM, Johnson S, Johns A. Randomized trial of a dissonance-based transdiagnostic group treatment for eating disorders: An evaluation of target engagement. J Consult Clin Psychol. 2019 Sep;87(9):772-786. doi: 10.1037/ccp0000430. PMID 31403814
- [Result] Stice E, Yokum S, Rohde P, Gau J, Shaw H. Evidence that a novel transdiagnostic eating disorder treatment reduces reward region response to the thin beauty ideal and high-calorie binge foods. Psychol Med. 2023 Apr;53(6):2252-2262. doi: 10.1017/S0033291721004049. Epub 2021 Oct 12. PMID 34635191
- [Derived] Stice E, Yokum S. Elevated reward, emotion, and memory region response to thin models predicts eating disorder symptom persistence: A prospective functional magnetic resonance imaging study. J Psychopathol Clin Sci. 2023 Aug;132(6):716-724. doi: 10.1037/abn0000843. PMID 37486363
- [Derived] Yokum S, Bohon C, Berkman E, Stice E. Test-retest reliability of functional MRI food receipt, anticipated receipt, and picture tasks. Am J Clin Nutr. 2021 Aug 2;114(2):764-779. doi: 10.1093/ajcn/nqab096. PMID 33851199

DOCUMENTS (1):
  • Informed Consent Form (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT03261050/ICF_000.pdf